CLINICAL TRIAL: NCT05780684
Title: Adaptive, Individualized Dose Escalation of Fluorouracil-Based Chemotherapy for Gastrointestinal Cancer: Pilot Study of the FOX Regimen
Brief Title: Individualized Dose Escalation of 5-FU for Gastrointestinal Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Gabriel A. Brooks, Associate Professor of Medicine, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY02001873; 22BRO873 (Other: Dartmouth Health)
Record Dates: First submitted 2023-03-10; First posted 2023-03-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Colorectal Cancer; Esophagus Cancer; Appendix Cancer; Small Bowel Cancer; Ampullary Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Esophageal Neoplasms; Appendiceal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Study Arm (Experimental): All patients in this single-study arm will be exposed to the FOX regimen, an adaptively dose-escalated chemotherapy regimen. The FOX regimen is comprised of oxaliplatin 85 mg/m2 IV on Day 1; leucovorin calcium 350 mg IV on Day 1; and infusional 5-FU IV over 46 hours (Days 1 and 2) - starting at a dose of 2,400 mg/m2 and adaptively adjusted toward a maximum dose of 3,200 mg/m2 over Cycles 2-4 using a clinical algorithm.
  Interventions: Other: FOX dose-escalation algorithm

INTERVENTIONS:
Other: FOX dose-escalation algorithm — Chemotherapy dose-escalation algorithm based on the FOLFOX and FOLFOXIRI regimens

SUMMARY:
This is a single-arm clinical trial to evaluate the feasibility of a chemotherapy regimen using adaptive, individualized dose escalation of 5-FU chemotherapy for patients who have good tolerance of the initial dose. Study participants will also receive oxaliplatin chemotherapy together with 5-FU, at standard doses. The goal of the study is to examine the feasibility and effectiveness of this approach, using individualized dose escalation of 5-FU in patients who do not have serious side effects at lower doses.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosis of metastatic or locally advanced/inoperable colorectal cancer or non-colorectal gastrointestinal cancer (including cancers of the stomach, esophagus, appendix, small bowel, and ampulla)
* Clinically appropriate staging imaging of the chest, abdomen, and pelvis performed within 30 days prior to registration
* ECOG Performance Status: 0-1

Exclusion Criteria:

* Any prior receipt of oxaliplatin or fluoropyrimidine chemotherapy (other than radiation-sensitizing fluoropyrimidine chemotherapy)
* Prior receipt of systemic chemotherapy in the 6 months prior to Day 1 of Cycle 1 of FOX (other than radiation-sensitizing chemotherapy)
* Known mismatch repair deficiency or microsatellite instability-high disease
* Known dihydropyrimidine dehydrogenase (DPD) deficiency, as identified by clinically indicated screening
* Any confirmed second malignancy that is likely to require systemic therapy during the course of the six-month study period, in the opinion of the enrolling investigator
* Any of the following baseline laboratory abnormalities:

  * Absolute neutrophil count (ANC) < 2,500/mm3
  * Platelet count < 100,000/mm3
  * Hemoglobin < 9 g/dL
  * Creatinine > 1.5 x ULN
  * Total bilirubin > 1.5 x ULN
  * AST/ALT > 5 x ULN
  * Patients who are unable to provide informed consent
  * Patients who are pregnant or breastfeeding
  * Patients who are incarcerated, homeless, or have active substance use disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-07-14 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients that receive dose intensified infusional 5-FU in Cycle 6 of the FOX regimen | Through day 1 of Cycle 6 of FOX regimen (cycle length is 14 days)
  The proportion of patients who receive dose-intensified infusional 5-FU (dosed at greater than or equal to 2,800 mg/m2) in Cycle 6 of the FOX regimen.

SECONDARY OUTCOMES:
Response rate to chemotherapy | Through 6 months from Cycle 1 Day 1 of FOX regimen
  Response rate (stratified by colorectal cancer vs. gastroesophageal cancer) as defined using RECIST 1.1 imaging criteria
Progression-free survival | Through 12 months from Cycle 1 Day 1 of FOX regimen
  Progression-free survival (PFS, stratified by colorectal cancer vs. gastroesophageal cancer, determined by retrospective review of medical records)
Dose intensity of 5-FU and oxaliplatin | Through day 1 of Cycle 6 of FOX regimen (cycle length is 14 days)
  Dose intensity of 5-FU and oxaliplatin over Cycles 1-6. Dose intensity will be calculated separately for each component of the FOLFOX regimen (5-FU infusion and oxaliplatin).
Mean plasma uracil concentration | Single treatment visit 0-30 days before Day 1 of Cycle 1 of FOX regimen, (cycle length is 14 days)
  Difference in mean plasma uracil concentration between patients who did and did not achieve sustained 5-FU dose escalation to ≥ 2,800 mg/m2 (primary endpoint)
5-FU drug exposure | Single treatment visit on Day 3 of treament Cycle 5 or Cycle 6 of FOX regimen, (cycle length is 14 days)
  5-FU drug exposure, measured as the area under the drug concentration curve (AUC). AUC will be calculated by multiplying the measured 5-FU concentration at steady state by the 5-FU infusion duration in hours.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel A Brooks, M.D., Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No